CLINICAL TRIAL: NCT06883968
Title: Effectiveness of a Therapeutic Physical Exercise Program During Outpatient Hospital Hemodialysis Treatment for the Improvement of Physical Capacity of Patients with Chronic Kidney Disease: a Randomized Controlled Multiple Cohort Clinical Trial
Brief Title: Therapeutic Exercise Programme to Improve the Functional Capacities, Depression and Anxiety of Patients with Chronic Kidney Disease During Haemodialysis Sessions.
Acronym: Actyren-HD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Responsible Party: Principal Investigator, Cristina Font, PhD in Comprehensive care and health services, University of Vic - Central University of Catalonia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACTYREN-01
Record Dates: First submitted 2025-02-18; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Exercise Therapy; Chronical Kidney Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic exercise intervention (Experimental): This group recibe one intervention demonstrated by a physiotherapist about therapeutic exercise to apply during hemodialysis session
  Interventions: Behavioral: Therapeutic exercise during hemodialysis session
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Therapeutic exercise during hemodialysis session — Participants in the intervention group will receive a therapeutic exercise program during hemodialysis sessions at the hospital. The physiotherapist, after assessing the participant, will plan a program with the sets and number of repetitions for the prescribed exercises based on the participant's condition.
  In this exercise program, the lower and upper extremities will be worked on with the aim of improving strength, balance, as well as contributing to the improvement of the participant's quality of life and mood.
  Arms: Therapeutic exercise intervention

SUMMARY:
Therapeutic Exercise During Outpatient Hemodialysis Treatment for Patients with Chronic Kidney Disease

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Treated for a minimum of 3 months with HD
* With clinical stability (good tolerance to sessions expressed as stable vital signs during the session)
* Voluntarily and with prior signed informed consent, have agreed to participate in the study

Exclusion Criteria:

* Physical or cognitive limitations that prevent following the intervention program
* Cardiovascular problems (unstable angina, uncontrolled arrhythmia, decompensated heart failure, pericarditis or myocarditis, severe untreated mitral or aortic stenosis)
* Uncontrolled arterial hypertension (SBP > 200 mmHg and DBP > 120 mmHg)
* Uncontrolled diabetes
* Severe neuropathies
* Acute systemic infection
* Severe renal osteodystrophy
* Stroke (cerebrovascular accident, transient ischemic attack)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2025-06-27 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Pre-intervention (A0) Post-intervention, after 16 weeks (A1) Up to 32 weeks (A2) Through study completion, an average of 1 year (A3)
  Physical capacity will be assessed using the Short Physical Performance Battery (SPPB) . The SPPB includes tests for balance, walking, and chair rise and sit.
  For the balance test, participants must stand in three positions: feet together, semi-tandem, and tandem. To earn 1 point and proceed to the semi-tandem position, they must remain with their feet together for at least 10 seconds. The same procedure applies for the tandem position.
  The walking test involves walking 4 meters at a comfortable pace, with the option of using assistive devices if necessary. The test is repeated twice, and the fastest time is selected. The scoring system is: 4 points for less than 4.82 seconds; 3 points for 4.48-6.20 seconds; 2 points for 6.21-8.70 seconds; 1 point for more than 8.70 seconds; and 0 points if the test is not completed.
  For the chair rise and sit test, participants must stand up and sit down 5 times as quickly as possible with arms crossed. The scoring is: 4 points for under 11.1

SECONDARY OUTCOMES:
Euro Quality of Life - EQ-5D-5L | Pre-intervention (A0) Post-intervention, after 16 weeks (A1) Up to 32 weeks (A2) Through study completion, an average of 1 year (A3)
  Quality of life will be assessed using the Euro Quality of Life - EQ-5D-5L questionnaire . This is a self-administered questionnaire consisting of two pages: the EQ-5D-5L descriptive system and the EQ Visual Analogue Scale. The descriptive system includes 5 dimensions (mobility, self-care, daily activities, pain/discomfort, anxiety/depression), and each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. To complete the questionnaire, the patient is asked to indicate their health status by marking the box that corresponds to the most appropriate level for each of the 5 dimensions. This results in a single-digit number, and when combined across the 5 dimensions, it forms a 5-digit number that describes the patient's health status. The EQ Visual Analogue Scale records the patient's perceived health status on a 20 cm vertical analogue scale. This information can be used quantitatively.
Barthel Index | Pre-intervention (A0) Post-intervention, after 16 weeks (A1) Up to 32 weeks (A2) Through study completion, an average of 1 year (A3)
  Functional independence during activities of daily living will be assessed using the Barthel Index. The Barthel Index is a 10-item scale. Each item assesses whether the patient is able to perform a task independently (2 points), with some assistance (1 point), or is unable to perform the task independently (0 points). The score for each item is summed, and the total is multiplied by 5 to convert it into a score ranging from 0 to 100. The higher the score, the greater the functional independence during activities of daily living .
HandGrip strength | Pre-intervention (A0) Post-intervention, after 16 weeks (A1) Up to 32 weeks (A2) Through study completion, an average of 1 year (A3)
  Handgrip strength of the dominant hand will be measured using the Jamar Hand Dynamometer (Sammons Preston, Inc, Molingbrook, IL) . The dominant hand will be determined according to the lateral preference inventory . The measurement will be taken with the participants seated in an upright position, with the arm to be used unsupported and parallel to the body. The grip width of the dynamometer will be adjusted to fit the size of each participant's hand so that the middle phalanges are placed on the inside of the handle. Participants will be asked to exert maximum force, starting with a submaximal trial to familiarize them with the testing procedure. The hand dynamometer has an intraclass correlation coefficient of 0.99 .
Hospital Anxiety and Depression Scale (HADS) | Pre-intervention (A0) Post-intervention, after 16 weeks (A1) Up to 32 weeks (A2) Through study completion, an average of 1 year (A3)
  Symptoms of anxiety and depression will be assessed using the Spanish version of the self-administered Hospital Anxiety and Depression Scale (HADS). The HADS consists of 14 items that assess the possible presence of depression and anxiety states in patients attending a non-psychiatric outpatient healthcare center. The HADS includes the anxiety and depression subscales, each consisting of 7 items scored using a 4-point Likert scale (e.g., [0] as usual, [1] not quite, [2] just a little, [3] never), giving a total score of 21 points for each subscale. This tool is validated for the Spanish population and has shown excellent internal consistency for its total score (alpha coefficient = 0.90), and moderate internal consistency for the anxiety (0.85) and depression (0.84) subscales .

OTHER OUTCOMES:
Age | Pre-intervention (A0)
  Age in years
Sex | Pre-intervention (A0)
  male or female
Location of the vascular access | Pre-intervention (A0)
  location of the vascular access in right or letf arm, or catheter
Duration of treatment with HD | Pre-intervention (A0)
  The time in years and months that the patient has been undergoing hemodialysis treatment
Charlson Comorbidity Index | Pre-intervention (A0)
  Screening for comorbidities
Weight | Pre-intervention (A0)
  weight in kilograms
Height | Pre-intervention (A0)
  height in meters
BMI | Pre-intervention (A0)
  weight and height will be combined to report BMI in kg/m^2
Smoking | Pre-intervention (A0)
  Smoker: Yes or No
Alcholism | Pre-intervention (A0)
  Consumes alcohol regularly: Yes or No

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Social Sciences and Community Health. Research Group on Methodology, Methods, Models and Outcomes of Health and Social Sciences . Faculty of Health Sciences and Welfare. University of Vic-Central of Catalonia, Vic 08500, Spain, Vic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
In the event that we decide to share the study data with other researchers, this will be done while maintaining anonymity or with additional consent from the participants.